CLINICAL TRIAL: NCT01300910
Title: Comparison of the Shang Ring With Conventional Surgical Methods: A Randomized Controlled Trial
Brief Title: Comparison of the Shang Ring With Conventional Surgical Methods
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: EngenderHealth (Other); Weill Medical College of Cornell University (Other); Kenya National AIDS & STI Control Programme (Other); Ministry of Medical Services, Kenya (Other); University Teaching Hospital, Lusaka, Zambia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10220
Record Dates: First submitted 2010-09-07; First posted 2011-02-23 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Circumcision, Male
Keywords: Adult Males; Circumcision; HIV prevention; Device; Shang Ring
MeSH Terms: interventions — Circumcision, Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): One group of men will undergo a circumcision using the Shang Ring and men are to return for regular follow-up visits to evaluate pain and wound healing. . The Shang Ring will be removed at 7 days, and the last scheduled follow-up visit is at 60 days.
  Interventions: Device: Shang Ring
- 2 (Active Comparator): One group of men will undergo a conventional circumcision using a WHO recommended surgical technique, either the forceps-guided method or the dorsal slit method. Men are to return for regular follow-up visits to evaluate pain and wound healing, with the last scheduled follow-up visit at 60 days.
  Interventions: Procedure: Male circumcision

INTERVENTIONS:
Device: Shang Ring — The Shang Ring is a sterile device consisting of two concentric medical grade plastic rings: an inner ring with a silicone band and an outer, hinged ring. The inner ring fits inside the outer ring which will lock when snapped together. The Shang Ring comes in multiple sizes. The appropriate size is determined through use of a measuring strip. To ensure that men cannot remove the device prematurely, the locking mechanism must be broken open using a tool that is similar to a scalpel handle. Then, a pair of special scissors, specifically designed for this purpose, is used to remove the inner ring after healing
  Arms: 1
Procedure: Male circumcision — A conventional surgical procedure will be performed, per WHO recommendations, involving: drawing a line to mark the amount of foreskin to be cut; cutting off the foreskin; hemostasis; and wound closure with sutures.
  Arms: 2

SUMMARY:
This is a randomized control trial of 400 adult male circumcision procedures with a one to one ratio between Shang Ring and the in-country standard surgical technique (forceps guided in Kenya and dorsal slit in Zambia).

DETAILED DESCRIPTION:
A randomized control trial of 400 adult male circumcision procedures with a one to one ratio between Shang Ring and the in-country standard surgical technique (forceps guided in Kenya and dorsal slit in Zambia)

Population: 400 men (200 at each site), HIV sero-negative men, ages 18-54, living in/around the two clinic sites seeking adult male circumcision

Duration: 2-4 months of recruitment; 60 days follow-up per participant; total expected duration of approximately 6 months in the field

Primary Objectives: (1) Compare the pain and acceptability of the Shang Ring procedure with the forceps guided surgical circumcision technique (Kenya) and the dorsal slit technique (Zambia) (2) Compare the safety and the course of wound healing, including the time to complete healing, between the Shang Ring adult male circumcision procedure and the standard surgical circumcision procedures (forceps guided in Kenya & dorsal slit in Zambia); (3) Compare the ease of the Shang Ring method versus standard circumcision surgical procedures

Primary Endpoints: (1) To compare the pain & acceptability of the circumcision methods, we will evaluate the following: post-operative pain; time to return to normal activity; patients' opinions of the Shang Ring and conventional procedures, and satisfaction with cosmetic results.

(2) To compare safety between methodologies, we will clinically compare and evaluate related adverse events and their severity. We will also compare the time to complete wound healing for each method. Complete wound healing is defined as no scab and dry skin by clinical assessment.

(3) We will evaluate the ease of surgery based on the duration of surgery and surgeons' opinions.

ELIGIBILITY:
Inclusion Criteria:

* Must be aged 18 and 54 years;
* Must be uncircumcised (on examination);
* Must be in good general health;
* Must be HIV sero-negative, with documentation of testing no more than one week before the procedure;
* Must be free of genital ulcerations or other visible signs of STI (on examination);
* Must be able to understand study procedures and requirements of study participation;
* Must agree to return to the healthcare facility for the full schedule of follow-up visits after his circumcision;
* Must freely consent to participate in the study and sign a written informed consent form;
* Must have a cell phone or access to a cell phone; and,
* Must agree to provide the study staff with an address, phone number, or other locator information while participating in the research study.

Exclusion Criteria:

* Has a known allergy or sensitivity to lidocaine or other local anesthesia;
* Takes a medication that would be a contraindication for elective surgery, such as an anticoagulant or steroid;
* Has known bleeding/clotting disorder (e.g. hemophilia); or
* Has an active genital infection, anatomic abnormality or other condition (e.g. severe obesity, diabetes or sickle cell anemia), which in the opinion of the surgeon, prevents the man from undergoing a circumcision as part of this study;
* Is not currently participating in another biomedical study.

Ages: 18 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Pain scores on the Visual Analog Scale | Within the first 48 hours after circumcision
  We will ask participants about pain they experienced during and soon after the procedure, and during the recovery period.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Up to six weeks after surgery
  We will classify circumcision-related adverse events, using the detailed definitions of moderate and severe events per standardized protocol definitions, based on WHO recommendations. Most post-operative complications are apparent within six weeks of surgery.

SECONDARY OUTCOMES:
Compare the cost of the Shang Ring procedure versus conventional surgery | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Marc Goldstein, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- Homa Bay District Hospital male circumcision clinic, Homa Bay, Nyanza, Kenya
- Society for Family Planning Clinic, Lusaka, Zambia

REFERENCES:
- [Derived] Hohlfeld A, Ebrahim S, Shaik MZ, Kredo T. Circumcision devices versus standard surgical techniques in adolescent and adult male circumcisions. Cochrane Database Syst Rev. 2021 Mar 31;3(3):CD012250. doi: 10.1002/14651858.CD012250.pub2. PMID 33786810